CLINICAL TRIAL: NCT04759547
Title: Handheld Ultrasound-assisted Versus Palpation-guided Labor Combined Spinal-epidural Analgesia: a Randomized Controlled Trial
Brief Title: Handheld Ultrasound-assisted Versus Palpation-guided Labor Combined Spinal-epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Kyung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2101-016-1186
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Labor Analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handheld ultrasound-assisted technique (Experimental): Participants will be received labor combined epidural-spinal analgesia using handheld ultrasound
  Interventions: Device: handheld ultrasound-assisted technique
- Conventional palpation-guided technique (Active Comparator): Participants will be received labor combined epidural-spinal analgesia using conventional landmark-guided technique
  Interventions: Other: conventional palpation-guided technique

INTERVENTIONS:
Device: handheld ultrasound-assisted technique — Ultrasound with 3D navigation function is used to determine the needle insertion point and the insertion angle.
  Arms: Handheld ultrasound-assisted technique
Other: conventional palpation-guided technique — The interspinous space is detected by palpation
  Arms: Conventional palpation-guided technique

SUMMARY:
Parturients who need combined spinal-epidural analgesia for labour analgesia are randomly assigned to two groups. For the handheld ultrasound-assisted technique group, ultrasound with 3D navigation function is used to determine the needle insertion point and the insertion angle. For the conventional palpation-guided technique group, the interspinous space is detected by palpation. Procedure time, the number of needle passes, the number of needle insertion attempts, success rate, and complications are compared.

DETAILED DESCRIPTION:
This study aims to determine whether handheld ultrasound-guidance can reduce procedural time for labor combined spinal-epidural analgesia compared with conventional surface landmark-guided technique.

ELIGIBILITY:
Inclusion Criteria:

- Adult parturients with ASA physical status classification I, II or III requiring a combined spinal-epidural for labor analgesia

Exclusion Criteria:

* Contraindication to neuraxial anesthesia (local anesthetics hypersensitivity, coagulopathy, needle insertion site infection, etc.)
* Difficulty in communication
* Severe cardiac disease
* History of spine surgery
* Anatomical abnormality of the lumbar spine
* Age under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Total duration of combined spinal-epidural procedure | During procedure
  Identifying time (time required to complete the preprocedural spinal ultrasound or the assessment by palpation) + Procedural duration (time from the initial Tuohy needle insertion through the skin to the completion of the threading of the epidural catheter)

SECONDARY OUTCOMES:
Number of passes | During procedure
  Number of times the puncture needle was redirected without removing it from the skin
Number of needle insertion attempts | During procedure
  Number of times the puncture needle was removed from the skin and reinserted
Procedural duration | During procedure
  time from the initial Tuohy needle insertion through the skin to the completion of the threading of the epidural catheter
Identifying time | During procedure
  time required to complete the preprocedural spinal ultrasound or the assessment by palpation
Success rate at the first needle pass | During procedure
  Success rate at the first needle pass
Success rate at the first attempt | During procedure
  Success rate at the first attempt
Need to use alternative methods | During procedure
  Need to use alternative methods for success
Number of interspace levels at which the insertion was attempted | During procedure
  Number of interspace levels at which the insertion was attempted
Success rate of dural puncture with needle-through-needle technique | During procedure
  Success rate of dural puncture with needle-through-needle technique
Incidence of radicular pain, paresthesia, and bloody tapping | During procedure
  Incidence of radicular pain, paresthesia, and bloody tapping during the procedure
Procedural pain using 11-point verbal rating scale | During procedure
  Degree of pain during the procedure using 11-point verbal rating scale (0=no pain, 10=most pain imaginable)
Procedural discomfort using 11-point verbal rating scale | During procedure
  Degree of discomfort during the procedure using 11-point verbal rating scale (0=no discomfort, 10=most discomfort imaginable)
Depth by ultrasound | During procedure
  Depth to the ligamentum flavum-dura mater complex (LFD) as determined by ultrasound
Actual needle depth (cm) | During procedure
  Depth of the needle when the epidural space and dural space are found (cm)
Failure of labor analgesia | Within 2 hours after the procedure
  The need to reinsert a new epidural catheter due to lack of sufficient analgesia within 2 hours of the primary insertion
Patient satisfaction using 11-point verbal rating scale | From the end of the procedure to delivery
  Patient satisfaction with the quality of labor analgesia using 11-point verbal rating scale (0=very unsatisfied, 10=very satisfied)
Incidence of inadvertent dural puncture | During procedure
  Incidence of inadvertent dural puncture
Incidence of postdural puncture headache | Up to 2 weeks
  Incidence of postdural puncture headache
Incidence of back pain postpartum at the site of epidural insertion | Up to 2 weeks
  Incidence of back pain postpartum at the site of epidural insertion

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Kyung Park, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simmons SW, Taghizadeh N, Dennis AT, Hughes D, Cyna AM. Combined spinal-epidural versus epidural analgesia in labour. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003401. doi: 10.1002/14651858.CD003401.pub3. PMID 23076897
- [Background] Neal JM, Brull R, Horn JL, Liu SS, McCartney CJ, Perlas A, Salinas FV, Tsui BC. The Second American Society of Regional Anesthesia and Pain Medicine Evidence-Based Medicine Assessment of Ultrasound-Guided Regional Anesthesia: Executive Summary. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):181-94. doi: 10.1097/AAP.0000000000000331. PMID 26695878
- [Background] Perlas A, Chaparro LE, Chin KJ. Lumbar Neuraxial Ultrasound for Spinal and Epidural Anesthesia: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):251-60. doi: 10.1097/AAP.0000000000000184. PMID 25493689
- [Background] Yoo S, Kim Y, Park SK, Ji SH, Kim JT. Ultrasonography for lumbar neuraxial block. Anesth Pain Med (Seoul). 2020 Oct 30;15(4):397-408. doi: 10.17085/apm.20065. PMID 33329842
- [Background] Park SK, Bae J, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Ultrasound-Assisted Versus Landmark-Guided Spinal Anesthesia in Patients With Abnormal Spinal Anatomy: A Randomized Controlled Trial. Anesth Analg. 2020 Mar;130(3):787-795. doi: 10.1213/ANE.0000000000004600. PMID 31880632
- [Background] Park SK, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Ultrasound-assisted vs. landmark-guided paramedian spinal anaesthesia in the elderly: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):763-771. doi: 10.1097/EJA.0000000000001029. PMID 31188153
- [Background] Bae J, Park SK, Yoo S, Lim YJ, Kim JT. Influence of age, laterality, patient position, and spinal level on the interlamina space for spinal puncture. Reg Anesth Pain Med. 2019 Nov 4:rapm-2019-100980. doi: 10.1136/rapm-2019-100980. Online ahead of print. PMID 31690644
- [Background] Tawfik MM, Atallah MM, Elkharboutly WS, Allakkany NS, Abdelkhalek M. Does Preprocedural Ultrasound Increase the First-Pass Success Rate of Epidural Catheterization Before Cesarean Delivery? A Randomized Controlled Trial. Anesth Analg. 2017 Mar;124(3):851-856. doi: 10.1213/ANE.0000000000001325. PMID 27183373
- [Background] Chin A, Crooke B, Heywood L, Brijball R, Pelecanos AM, Abeypala W. A randomised controlled trial comparing needle movements during combined spinal-epidural anaesthesia with and without ultrasound assistance. Anaesthesia. 2018 Apr;73(4):466-473. doi: 10.1111/anae.14206. Epub 2018 Jan 10. PMID 29322504
- [Background] Arzola C, Mikhael R, Margarido C, Carvalho JC. Spinal ultrasound versus palpation for epidural catheter insertion in labour: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jul;32(7):499-505. doi: 10.1097/EJA.0000000000000119. PMID 25036283
- [Derived] Bae J, Kim Y, Yoo S, Kim JT, Park SK. Handheld ultrasound-assisted versus palpation-guided combined spinal-epidural for labor analgesia: a randomized controlled trial. Sci Rep. 2023 Dec 27;13(1):23009. doi: 10.1038/s41598-023-50407-7. PMID 38155223